CLINICAL TRIAL: NCT01029678
Title: Phase II Study Evaluating Treatment With Oral Navelbine and Cisplatin Administered Weekly and Concomitant Radiotherapy in Elderly Patients With no Operable NSCLC
Brief Title: Concomitant Radio-chemotherapy in the Elderly
Acronym: RACCOSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Pierre Fabre Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I08011
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Locally advanced lung cancer; Elderly patients; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- experimental (Experimental)
  Interventions: Drug: Cisplatin IV; Drug: Vinorelbine; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cisplatin IV — Cisplatin IV 30 mg/m2/ (Day 1, Day 8, Day 15, Day 22, Day 29, Day 36)
Drug: Vinorelbine — Vinorelbine per os 30 mg/m2/(day1, day8, day15, day22, day29, day36
Radiation: Radiotherapy — 66Gy, 33 fractions, 6 week

SUMMARY:
The purpose of this study is to evaluate the safety of non small cell lung cancer (NSCLC) treatment with cisplatin and oral vinorelbine administered weekly associated with concomitant radiotherapy in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Independent patients (based on the score of geriatric frailty: IADL = 0, ADL = 0, no geriatric syndrome, low comorbidity (comorbidity index of Charlson to 3 or 4), depression score 0-1)
* Performance Status (ECOG) ≤ 1
* Weight loss <10% of usual weight in the last 3 months
* Life expectancy greater than 12 weeks
* Hematologic function: neutrophils> 1.5 x 10**9 / l, hemoglobin> 9.5 g / dl, platelets > 100 x 10**9 / l)
* Renal function: creatinine clearance ≥ 50 ml / min calculated by the formula of MDRD
* Normal liver function: bilirubin < Limit of Normal (ULN), SGOT and / or SGPT <2.5 x UNL
* Respiratory Function: FEV ≥ 40% predicted, PaO2 ≥ 60 mm Hg, KCO ≥ 60% predicted
* Patient affiliated to a social security regimen or beneficiary of such regimen
* Informed consent signed

The disease

* Pathological anatomy: CBP non-small cell (squamous cell carcinoma, adenocarcinoma, large cell carcinoma, undifferentiated carcinoma) histologically or cytologically proven
* Stage IIIAN2 considered inoperable stage IIIB
* Presence of at least one measurable target
* Delay at least three weeks between surgery and initiation of treatment
* No prior treatment with chemotherapy or radiotherapy for lung cancer

Exclusion Criteria:

* Age < 70 years
* Performance Status (ECOG) ≥ 2
* Hematologic function: neutrophils <1.5 x 10**9 / l, hemoglobin <9.5 g / dl, platelets <100 x 10**9 / l)
* Renal function: creatinine clearance <50 ml / min calculated by the formula of MDRD
* Hepatic: bilirubin> Upper Limit of Normal (ULN), SGOT and / or SGPT> 2.5 x ULN
* Respiratory Function: FEV <40% predicted, KCO <60% predicted, PaO2 <60 mmHg
* Peripheral neuropathy grade> 1
* Unstable cardiac pathology requiring treatment (heart failure, angor of effort, arrhythmia) or previous myocardial infarction older than 12 months
* Deafness not paired or deafness requiring major achievement of an audiogram-cons may indicate taking cisplatin
* Neurological or psychiatric disorders prohibiting the understanding of the test
* Previous history of cancer except basal cell cancer, carcinoma in situ of the cervix treated or any other cancer treated with surgery alone or radiotherapy alone extra-thoracic recurrence-free 5 years
* Significant malabsorption syndrome or disease affecting the functioning of the gastrointestinal tract

The disease

* Pathological anatomy: Bronchioloalveolar carcinoma, neuroendocrine carcinoma, small cell carcinoma
* Metastatic disease
* Pleural drain
* Carcinomatous lymphangitis
* Operable Cancer
* Previously treated for lung cancer disease: radiotherapy, chemotherapy, hormonal therapy, endobronchial suctioning older less than eight days

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Acute toxicity | during treatment and during the 4 weeks following the end of treatment

SECONDARY OUTCOMES:
Late toxicity | 6 months after the end of the treatment
Overall response rate | 4 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chrystèle LOCHER, MD, Study Chair — CH Meaux
Locations (5):
- France (5):
  - CHU Brest, Brest
  - Centre Hospitalier GAP, Gap
  - Département de Pathologie Respiratoire du CHU de Limoges, Limoges
  - CH de Meaux, Meaux
  - CHU Reims, Reims